CLINICAL TRIAL: NCT01106976
Title: Imaging Biomarkers of Progression of Mobility Impairment in Parkinson Disease
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Other Study IDs: E7285-R
Record Dates: First submitted 2010-04-14; First posted 2010-04-20 (Estimated); Results first posted 2016-02-01 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2015-12

CONDITIONS: Parkinson's Disease
Keywords: PET; acetylcholine
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1 Parkinson disease subjects: Subjects with Parkinson disease who previously participate in a motor and brain PET (brain positron emission tomography) imaging study who were invited for a longitudinal observational study.

SUMMARY:
The purpose of this research is to evaluate changes in cholinergic brain activity over time in subjects with Parkinson disease.

DETAILED DESCRIPTION:
The project will apply positron emission tomography (PET) of acetylcholinesterase to study non-dopaminergic (i.e. cholinergic) brain changes over time in subjects with Parkinson disease. Acetylcholinesterase PET imaging was used to assess cholinergic changes over time in this study. Acetylcholinesterase PET imaging is a diagnostic test as the investigator does not assign specific interventions to the subjects of the study based on the acetylcholinesterase PET. Therefore, this is an observational study as defined as following: studies in human beings in which biomedical and/or health outcomes are assessed in pre-defined groups of individuals. Subjects in the study may receive diagnostic, therapeutic, or other interventions, but the investigator does not assign specific interventions to the subjects of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet the UK Parkinson's Disease Society Brain Bank Research Center clinical diagnostic criteria for PD.
* Hoehn and Yahr stages 1-2.5 at initial recruitment in baseline study.
* Absence of dementia confirmed by neuropsychological testing at initial recruitment in baseline study.

Exclusion Criteria:

* contra-indication for magnetic resonance study
* Pregnancy or breastfeeding

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recruited in previous study
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2010-05; Primary Completion 2014-09 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaas I Bohnen, MD PhD, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Bohnen NI, Frey KA, Studenski S, Kotagal V, Koeppe RA, Scott PJ, Albin RL, Muller ML. Gait speed in Parkinson disease correlates with cholinergic degeneration. Neurology. 2013 Oct 29;81(18):1611-6. doi: 10.1212/WNL.0b013e3182a9f558. Epub 2013 Sep 27. PMID 24078735
- [Result] Muller ML, Albin RL, Kotagal V, Koeppe RA, Scott PJ, Frey KA, Bohnen NI. Thalamic cholinergic innervation and postural sensory integration function in Parkinson's disease. Brain. 2013 Nov;136(Pt 11):3282-9. doi: 10.1093/brain/awt247. Epub 2013 Sep 20. PMID 24056537
- [Result] Kotagal V, Albin RL, Muller ML, Koeppe RA, Frey KA, Bohnen NI. Diabetes is associated with postural instability and gait difficulty in Parkinson disease. Parkinsonism Relat Disord. 2013 May;19(5):522-6. doi: 10.1016/j.parkreldis.2013.01.016. Epub 2013 Feb 23. PMID 23462483

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 67 patients with Parkinson disease
Pre-assignment Details: Patient with Parkinson disease with no contra-indication for MRI.
Groups:
- Group 1 Parkinson Disease Subjects: Prospective cohort study. 59 PD patients; Hoehn and Yahr stage 1-3) underwent [C-11]methyl-4-piperidinyl propionate (PMP) acetylcholinesterase (AChE) brain PET imaging at baseline and at 3-4 year follow-up. AChE PET imaging assesses cholinergic terminal integrity with cortical uptake reflecting largely basal forebrain neuron integrity and thalamic uptake principally reflecting pedunculopontine nucleus integrity.
Period: Overall Study
Arm/Group | Group 1 Parkinson Disease Subjects
Started | 67
Completed | 59
Not Completed | 8
Not completed — Lost to Follow-up | 8

BASELINE CHARACTERISTICS:
Population: Parkinson disease, minimum age of 50.
Groups:
- Group 1 Parkinson Disease Subjects: Prospective cohort study. 59 PD patients
Arm/Group | Group 1 Parkinson Disease Subjects
Number analyzed (Participants) | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.7 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 60
Region of Enrollment [Number; unit: participants]
  United States | 67

OUTCOME MEASURES:

1. Primary Outcome: AChE PET Neuroimaging
Description: AChE PMP PET hydrolysis rate outcome measure. AChE [11C]PMP hydrolysis rates (k3) were estimated using the striatal volume of interest (defined by manual tracing on the MRI scan of the putamen and caudate nucleus) as the tissue reference for the integral of the precursor delivery. This measure is a proxy measure for the count of cholinergic nerve terminals in the basal forebrain innervation the cortical mantle.
Time Frame: 4 yr
Population: Parkinson disease.
Measure: Mean (Standard Deviation); unit: 1/min
Groups:
- Parkinson Disease: Prospective cohort study of Parkinson disease subjects.
Arm/Group | Parkinson Disease
Number analyzed (Participants) | 59
1/min
  baseline forebrain cortical AChE activity | 0.0238 (0.0029)
  4-yr forebrain cortical AChE follow-up activity | 0.0226 (0.0032)
Statistical Analysis 1: Comparison: Parkinson Disease; Paired t-test. Hypothesis of significant cholinergic interval changes over the study interval period; Test type: Superiority or Other; p = 0.0009, t-test, 1 sided; Mean Difference (Net) = 0.0012

ADVERSE EVENTS:
Time Frame: 1.5-4 yr
Groups:
- Parkinson: Longitudinal cohort
Arm/Group | Parkinson
Serious Adverse Events (participants affected / at risk) | 0/67
Other Adverse Events (participants affected / at risk) | 1/67
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Parkinson (N=67)
scanner claustrophobia (Psychiatric disorders) | 1 (1) — expected mild AE

LIMITATIONS AND CAVEATS:
Observational study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No